CLINICAL TRIAL: NCT00000197
Title: Propranolol for Treatment of Cocaine Addiction
Brief Title: Propranolol for Treatment of Cocaine Addiction - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Kyle Kampman, University of Pennsylvania
Purpose: Treatment
Other Study IDs: NIDA-00238-2; K20DA000238 (NIH)
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Propranolol

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of propanolol in the early treatment of cocaine dependence.

ELIGIBILITY:
Please contact site for information.

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1987-01; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Side effects
Cocaine use
Cocaine withdrawal
Cocaine craving
Mood and anxiety
Clinical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Kampman, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States